CLINICAL TRIAL: NCT05918510
Title: Observational Study of Viral BIOmarkers and microRNAs in Tumors Orofarynx and Occult Tumors Positive for Papilloma Virus
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Istituto Clinico Humanitas (Other); Istituto Europeo di Oncologia (Other); Azienda Policlinico Umberto I (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); University of Firenze and Siena, Napoli, Italy (Other); Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Other Study IDs: RS1647/22
Record Dates: First submitted 2023-03-29; First posted 2023-06-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-06

CONDITIONS: Squamous Cell Carcinoma of the Oropharynx; Carcinomas of Unknown Primary Site; High-risk Human Papillomavirus Infection; Liquid Biopsy; Lymph Node Metastasis; Occult Tumor of the Head and Neck Area
Keywords: Oropharyngeal Tumor; Occult Cancer; HPV Infection; head-neck area
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphatic Metastasis; Oropharyngeal Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: High miR value
  Interventions: Diagnostic Test: Study of Viral BIOmarkers and microRNAs in Tumors Orofarynx
- Group 2: Control group
  Interventions: Diagnostic Test: Study of Viral BIOmarkers and microRNAs in Tumors Orofarynx

INTERVENTIONS:
Diagnostic Test: Study of Viral BIOmarkers and microRNAs in Tumors Orofarynx — The prospective observational study involves the collection of tissue, blood and saliva samples from OPSCC and occult T patients for detection of HPV-DNA/RNA, miRNA and mutation profile from DNA with centralized analysis of samples at IRCCS Regina Elena National Cancer Institute.

SUMMARY:
Based on the evidence summarized in the introduction, the clinician hypothesize that the detection of the presence and expression of HPV-DNA, certain miRNAs, and a certain mutational profile in the tissues and biological fluids of these patients, may have important prognostic and diagnostic value not only in HPV-related OPSCCs but also in HPV+ occult T. Accordingly, this study aims to aim to better characterize their potential as biomarkers and to detect the possibility of their their use to implement the sensitivity and specificity of radiological methodologies (PET-CT and MRI), already in use in clinical practice, for monitoring disease progression in this specific subgroup. Finally, by using the collected material to generate organoids and Patient Derived Xenograft (PDX), the study also aims to identify possible new molecular drugs, which could solve the problem of resistance to radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinomas of the oropharynx and occult neoplasms with lymph node metastases laterocervical cytologically positive for squamous cell carcinoma treated with TORS or RT or RT/CT
* Age > 18 years
* ECOG performance status <_ 2
* Ability to follow study procedures and complete questionnaires
* Signature of informed consent

Exclusion Criteria:

* Presence of distant metastases at the time of diagnosis
* Previous cancer of the head and neck district
* Second tumor in therapy or follow-up for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinomas of the oropharynx and occult neoplasms with lymph node metastases Cytologically positive laterocervical squamous cell carcinoma treated with TORS or RT or RT/CT
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-04-04 (Estimated); Study Completion 2029-04-04 (Estimated)

PRIMARY OUTCOMES:
Accouracy | Baseline
  Investigating the kinetics of HPV-DNA and miRNAs in patients with oropharyngeal and occult T tumors with laterocervical metastasis. Conducting this study will allow us to collect the information needed to be able to generate hypotheses and design a subsequent larger study.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided